CLINICAL TRIAL: NCT01019642
Title: Effect of Vitamin D Supplementation on C-reactive Protein and Insulin Resistance in Postmenopausal Women With Type 2 Diabetes Mellitus
Brief Title: Vitamin D, C-reactive Protein and Insulin Resistance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Collaborators: Instituto Mexicano del Seguro Social (Other Government); Ellison Medical / International Nutrition Foundation (Unknown); Tufts University (Other)
Responsible Party: Mario E. Flores, Instituto Nacional de Salud Publica
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 120-6371
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Diabetes; Low-intensity Chronic Inflammation; Insulin Resistance
Keywords: vitamin D; diabetes; C-reactive protein; insulin resistance
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Experimental): Cholecalciferol, 4,000 IU/d for 6 months
  Interventions: Drug: cholecalciferol
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: cholecalciferol — 4,000 IU per day during 6 months. Capsule form.
  Arms: Vitamin D
Drug: placebo — no active principles given.
  Arms: Placebo

SUMMARY:
Randomized, double blind, placebo-controlled clinical trial of vitamin D supplementation (cholecalciferol, 4,000 IU/day for 6 months, in 104 postmenopausal women with type 2 diabetes mellitus.

The objective was to evaluate the effect of vitamin D supplementation on C-reactive protein (CRP) and insulin resistance in women with type 2 diabetes mellitus (T2DM).

The trial was conducted from March to October 2008 at the Hospital of the Mexican Social Security in Cuernavaca, Mexico.

DETAILED DESCRIPTION:
Methods. Randomized, double blind, placebo-controlled clinical trial. We selected 104 postmenopausal women, ages 45 to 65, with uncomplicated T2DM and BMI ≥25. Women with history of kidney or liver disease, BMI>40, autoimmune disease or cancer were not included in the study.

Participants were randomly assigned to receive either a capsule containing 4,000 IU of vitamin D3 (cholecalciferol, n=52) or placebo (n=52), once a day during 6 months.

Outcome variables were serum CRP, measured with a high-sensitivity assay (nephelometry), and HOMA-IR. Serum vitamin D (25-OH-D) was measured by HPLC. Outcome variables were measured at baseline, and 3 and 6 months thereafter. All participants received diet and physical activity counseling, and visited the clinic for medical check-up once a month.

Baseline Results. Mean age was 56.8 ± 5.1 y. Baseline BMI was 30.7 ± 3.9. Median CRP concentration was 5.0 mg/L (Interquartile range: 1.0, 8.5). HOMA index at baseline was 7.13 ± 3.8. Serum 25-OH-D concentration at baseline was 54.5 ± 15.7 nmol/L (~22 ng/mL). Almost 94% of patients had baseline serum 25-OH-D levels <80 nmol/L, and 25% were below 40 nmol/L. No one had levels <20 nmol/L. There were no statistical differences on important variables by treatment group at the onset of study.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus w/ < 10 yrs of diagnosis
* Postmenopausal
* Overweight or obesity (BMI >=25)
* Treated with metformin

Exclusion Criteria:

* BMI >=40
* Liver or kidney disease
* Other important chronic disease: i.e. cancer, autoimmune.
* Receiving insulin

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2008-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Serum C-reactive protein concentrations, measured by a high-sensitivity assay -nephelometry-. | 3 and 6 months
Insulin resistance, measured by HOMA-IR index | 3 and 6 months

SECONDARY OUTCOMES:
Serum 25-OH-vitamin D3 levels | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mario E Flores, MD, MSc, Principal Investigator — Instituto Nacional de Salud Publica, Mexico
Locations (1):
- Instituto Mexicano del Seguro Social, Cuernavaca, Morelos, Mexico

REFERENCES:
- [Background] Flores M. A role of vitamin D in low-intensity chronic inflammation and insulin resistance in type 2 diabetes mellitus? Nutr Res Rev. 2005 Dec;18(2):175-82. doi: 10.1079/NRR2005104. PMID 19079903
- [Derived] Munoz-Aguirre P, Flores M, Macias N, Quezada AD, Denova-Gutierrez E, Salmeron J. The effect of vitamin D supplementation on serum lipids in postmenopausal women with diabetes: A randomized controlled trial. Clin Nutr. 2015 Oct;34(5):799-804. doi: 10.1016/j.clnu.2014.10.002. Epub 2014 Oct 13. PMID 25453396